CLINICAL TRIAL: NCT00622687
Title: Comparision Between Maximally Tolerated Intravenous Iloprost Doses Versus Low-Dosed Iloprost for a 21-Day Treatment Course
Brief Title: Effect of Different Iloprost Doses on Symptoms in Systemic Sclerosis
Acronym: ILODOSE
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: sufficient number to reach the primary endpoint and as planned
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Schering-Plough (Industry)
Responsible Party: Riemekasten, PD Dr. med., Cahrité Universitätsmedizin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILO-1998; Schering GmbH
Record Dates: First submitted 2008-02-14; First posted 2008-02-25 (Estimated); Last update posted 2008-02-25 (Estimated); Status verified 2007-12

CONDITIONS: Systemic Sclerosis
Keywords: iloprost; systemic sclerosis; digital ulcers; observational study; randomized
MeSH Terms: conditions — Scleroderma, Systemic; digital ulcers | interventions — Iloprost

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator): low dose iloprost therapy 0.5 ng/kg x min
  Interventions: Drug: iloprost low dose; Drug: iloprost therapy up to 2 ng/kg x min
- B (Active Comparator): high-dose therapy
  Interventions: Drug: iloprost; Drug: iloprost therapy up to 2 ng/kg x min

INTERVENTIONS:
Drug: iloprost — 0.5-2 ng/kg x min for 6hours a day for 21 consecutive days
  Other Names: intravenous ilomedin
  Arms: B
Drug: iloprost low dose — 0.5 ng/kg x min over 6 h per day for 21 consecutive days
  Other Names: intravenous ilomedin
  Arms: A
Drug: iloprost therapy up to 2 ng/kg x min — starting therapy at doses of 0.5 ng/kg x min, increase the dose every two days for 0.5 ng/kg x min up to the maximally tolerated dose or to 2 ng/kg x min
  Other Names: ilomedin treatment

SUMMARY:
This study compared the efficacy of different dosages of long-term iloprost treatment on Raynaud's phenomenon, ulcer healing, skin thickening, and progression of internal organ sclerosis in systemic sclerosis (SSc).

Methods. 50 SSc patients were 1:1 randomised either for maximally tolerated dose up to 2 ng/kg body weight [bw] per minute or low dose (0.5 ng/kg bw per minute) intravenous iloprost administration, for six hours daily over 21 days. The effect on RP, ulcer healing, skin thickness, oesophagus function, lung involvement as assessed by lung function parameters FVC and DLCO, and side effects were measured.

Conclusions. The efficacy of prolonged administration of iloprost is also achieved with low dose iloprost by long term treatment. The effects suggest a disease-modifying capability of iloprost, but further studies are needed to proof this hypothesis.

DETAILED DESCRIPTION:
50 SSc patients (23 patients with limited SSc; 15 patients with diffuse SSc, and 12 patients with overlap syndromes fulfilling the ACR criteria for systemic sclerosis) and suffering from severe Raynaud's phenomenon were included into the study after written informed consent to participate in this study. Severe Raynaud's phenomenon was defined by a high burden of disease, by trophic skin changes, or the presence of digital ulcers.

Patients suffering from SSc related RP and/or digital ulceration were randomized 1 : 1 to one of the following groups that received either high or low dose infusions of iloprost for 21 consecutive days given once or twice a year. High dose patients (n=25) started on 0.5ng per kg bw and min over 6 hours a day. Depending on the tolerability the dosages were increased in increments gradually every two days for 0.5 ng/kg x min. The maximum dose administered was 2.0ng/kg bw and min. Low dose patients (n=25) were permanently treated with 0.5ng/kg bw over 6 hours per day for 21 consecutive days.

ELIGIBILITY:
Inclusion Criteria:

* patients with secondary Raynaud's phenomenon suffering from severe Raynaud-'s phenomenon with trophical changes or from digital ulcers with written informed consent. Patients had to be stable for their systemic disease and were on stable medication concerning immunosuppression or vasoactive therapies for three months.

Exclusion Criteria:

* Current smokers, patients with a history of gastric ulcers in the last three months, a cardiac ejection fraction below 25%, patients with severe organ involvement or other uncontrolled diseases such as instable angina pectoris, severe anaemia, coagulopathies, azothaemia, cerebral stroke in the last 6 months or malignant diseases were excluded from the study. The last iloprost therapy had to be finished at least 6 months ago. Participation in other studies during the last 4 weeks was also not allowed. For fertile women, a negative pregnancy test was required.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 1997-09; Primary Completion 2003-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Healing of digital ulcers | 5 weeks

SECONDARY OUTCOMES:
Duration of RP | 6 weeks
Frequency of RP | 6 weeks
changes in lung function | 4 years
changes in MRSS | 6 years
subjective improvement of esophagus function | 1 year
subjective benefit from iloprost therapy | 1 year
side effecs | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Gabriela Riemekasten, MD, Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Charrité Universitätsmedizin, Berlin, State of Berlin, Germany

REFERENCES:
- [Background] Riemekasten G, Jepsen H, Burmester GR, Hiepe F. [Iloprost administration over 21 days as an effective therapy in systemic scleroderma--case report and review of the literature]. Z Rheumatol. 1998 Apr;57(2):118-24. doi: 10.1007/s003930050070. German. PMID 9627952
- [Derived] Kawald A, Burmester GR, Huscher D, Sunderkotter C, Riemekasten G. Low versus high-dose iloprost therapy over 21 days in patients with secondary Raynaud's phenomenon and systemic sclerosis: a randomized, open, single-center study. J Rheumatol. 2008 Sep;35(9):1830-7. Epub 2008 Jul 15. PMID 18634152
- See also: Related Info — http://www.charite.de
- See also: Related Info — http://www.Sklerodermie.info